CLINICAL TRIAL: NCT06577688
Title: Assessing the Feasibility of Classifying People Using a Machine-learning Approached Based on Features Derived From Smartphone Video Data Recorded at the Person's Fingertip
Brief Title: Smartphone Blood Pressure Measurement to Screen for Hypertension
Acronym: Optiscreen
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Patrick Schoettker, Professor, Centre Hospitalier Universitaire Vaudois
Other Study IDs: 2023-00851
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Blood Pressure; Blood Pressure Disorders
Keywords: blood pressure; smartphone; Home blood pressure monitoring; Blood pressure disorders screening

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Volunteer presumed healthy: People presumed healthy undergoing blood pressure measurement with a standard cuff device and with a Smartphone
  Interventions: Other: Blood pressure measurement
- Volunteer suspected of arterial hypertension: People addressed for a suspected diagnosis of arterial hypertension undergoing a home blood pressure monitoring and measurements with a smartphone
  Interventions: Other: Blood pressure measurement

INTERVENTIONS:
Other: Blood pressure measurement — Blood pressure measurement using a standard cuff device and a smartphone

SUMMARY:
The goal of this observational study is to assess the feasibility of classifying people whose blood pressures are within hypertensive range using a machine-learning approach based on features derived from smartphone video data recorded at the patient's fingertips. The main question[s] it aims to answer are:

Is a smartphone a reliable device for high blood pressure screening ? Is a smartphone a reliable device for blood pressure monitoring ? Participants will record their blood pressure with a smartphone at their fingertips and with an approved cuff device, 3 times in the morning and 3 times in the evening for 7 days. There will be two groups, a volunteer presumed healthy, and a volunteer addressed for a Home Blood pressure monitoring with the diagnosis of hypertension suspected.

Researchers will compare the two groups to see if the smartphone can be reliable in terms of diagnosis and monitoring of the blood pressure comparing to a standard cuff device.

DETAILED DESCRIPTION:
This is a single-center observational pilot study. Data will be collected prospectively on 100 participants (maximum of 120) with, ideally, 50 presumed healthy volunteers and 50 participants with a suspected diagnosis of hypertension. Presumably healthy volunteers will be recruited via flyers and participants presumed to be hypertensive will be recruited by the hypertension unit of the CHUV, where they are referred for the search for a diagnosis of hypertension.

To comply with the International Hypertension Societies guidelines for LMWH, participants will measure their blood pressure for 7 consecutive days, in the morning (before taking medications and food) and in the evening. (before dinner). At each measurement time point, participants will acquire three separate measurements, one minute apart. Participants will record signals by placing a fingertip of the right hand over a smartphone camera, while simultaneously acquiring a baseline blood pressure measurement using a validated cuff device (WatchBP O3 Ambulatory, Microlife, Widnau, Switzerland) on the left arm. Please note that the smartphone and armband will be provided by the site investigator. The data recorded using the smartphone will be processed and directly compared to the values obtained using the inflatable cuff device.

In accordance with international guidelines for LMWH (except those of the American Heart Association), the threshold for hypertension is set at systolic blood pressure values ≥ 135 mmHg and/or diastolic blood pressure values ≥ 85 mmHg.

The aim of this study is to evaluate the feasibility of classifying people whose blood pressure is in the hypertensive range or not, using a method based on machine learning. To do this, optical data will be recorded at the fingertip from a smartphone camera following the HBPM measurement protocol. The optical signals will then be processed by a machine learning method to obtain the classification. In other words, we will attempt to evaluate the reliability of the machine learning method compared to the automatic oscillometric brachial cuff and therefore evaluate the feasibility of using the smartphone as a potential future tool for diagnosis, screening and monitoring hypertension.

The methods of screening, diagnosis and monitoring of hypertensive pathologies are precise but require cumbersome equipment and are sometimes poorly available. We hypothesize that smartphones can be used because of to their availability and their capacity to generate quality optical signals, as a discriminating classifier in arterial hypertension thanks to the precision of a machine learning model hypothetically greater than a classification carried out by a random level.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature
* Men or women older than 18 years old
* Good understanding of written and oral speaking used at the center where the study will be carried out

Exclusion Criteria:

* Patients that cannot sign informed consent
* Patients in emergency situation, are not legally competent, cannot understand the situation or are vulnerable
* Unable to participate due to pain or stress [12]
* Known or suspected non-compliance (e.g. drug or alcohol abuse, language problems, psychological disorders, dementia)
* Patients older than 80 years old [4] [13]
* Known pregnancy
* Known unstable cardiac condition (myocardial infarction < 1 week, decompensated heart failure, pulmonary embolism)
* End-stage renal disease (GFR < 15/min/1.73m2 and/or dialysis) [4] [14] [15] [16]
* Diabetes mellitus [15] [8]
* Known (or assessed by recording heart rate and using pulse palpation, as recommended in ESC/ESH guidelines [1]) cardiac arrhythmia (atrial fibrillation, numerous extrasystoles and important bradycardia/bradyarrhythmia, bigeminy, trigeminy, isolated VPB) [4] [1] [7] [15] [17]
* SBP or DBP difference between two arms >10 mmHg [8] [18]
* Patient with finger lesions that would alter the correct capture of signals by the mobile phone.
* Known mobile phone contact dermatitis (caused by metal allergens, notably nickel and chromium
* Incapacity of properly using the smartphone (i.e. incapacity of obtaining a recording with sufficient signal quality after the dedicated training)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For this study, the aim is to reach balanced classes, with at least 40% of non-hypertensive patients and 40% of hypertensive patients. In order to approach such distributions, both healthy volunteers and patients suspected of hypertension visiting the CHUV Hypertensive Unit for diagnosis confirmation will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Reliability of smartphone's blood pressure measurements | 7 days
  Reliability of smartphone's blood pressure measurements to discriminate values within hypertension range compared to standard cuff device

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schoettker, PhD, Principal Investigator — Centre Hospitalier Universitaire Vaudois

IPD SHARING:
Plan to Share IPD: Undecided